CLINICAL TRIAL: NCT00510016
Title: Efficacy of Clonidine in the Treatment of Neonatal Abstinence Syndrome: A Prospective, Double Blind, Randomized Controlled Trial
Brief Title: Clonidine as Adjunct Therapy for the Treatment of Neonatal Abstinence Syndrome
Acronym: NAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21DA016288-01A1 (NIH); 1R21DA016288-01A1 (NIH)
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2007-07

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: infants; opioid withdrawal; abstinence syndrome; methadone; heroin
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clonidine treatment (Experimental): Infants intrauterine exposed to opioids (heroin or methadone) that demonstrate signs and symptoms of withdrawal with withdrawal scores (modified Finnegan score) greater than 9 on to consecutive scores taken 4 hours apart.
  Interventions: Drug: Clonidine HCL

INTERVENTIONS:
Drug: Clonidine HCL — Duraclon 1 microgram/kg every 4 hours given p.o. as per algorithm
  Other Names: Duraclon

SUMMARY:
To test the hypothesis that the combination of the tincture of opium (DTO) and clonidine will be more effective in treating infants with neonatal abstinence syndrome (opioid withdrawal) than tincture of opium (DTO) alone.

ELIGIBILITY:
* neonates born at gestational age of 35 weeks or greater
* neonates aged 0 to 14 days
* prenatally exposed to opioids
* severe NAS defined as 2 consecutive modified Finnegan Scores (MFS) > or = 9

Exclusion Criteria:

* < 35 weeks gestational age
* Intrauterine growth retardation defined as <5%tile of gestational age
* postnatal treatment with barbiturates or benzodiazepines,
* major congenital anomalies
* major concomitant medical illness requiring oxygen therapy, intravenous fluids or medications.
* breastfed infants

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2002-07; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Length of treatment for neonatal abstinence syndrome | duration of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Estelle B Gauda, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

REFERENCES:
- [Background] Hoder EL, Leckman JF, Poulsen J, Caruso KA, Ehrenkranz RA, Kleber HD, Cohen DJ. Clonidine treatment of neonatal narcotic abstinence syndrome. Psychiatry Res. 1984 Nov;13(3):243-51. doi: 10.1016/0165-1781(84)90039-8. PMID 6597462
- [Background] Gold MS, Pottash AL, Extein I, Kleber HD. Clonidine and opiate withdrawal. Lancet. 1980 Nov 15;2(8203):1078-9. doi: 10.1016/s0140-6736(80)92295-3. No abstract available. PMID 6107698
- [Derived] Agthe AG, Kim GR, Mathias KB, Hendrix CW, Chavez-Valdez R, Jansson L, Lewis TR, Yaster M, Gauda EB. Clonidine as an adjunct therapy to opioids for neonatal abstinence syndrome: a randomized, controlled trial. Pediatrics. 2009 May;123(5):e849-56. doi: 10.1542/peds.2008-0978. Epub 2009 Apr 27. PMID 19398463